CLINICAL TRIAL: NCT02227134
Title: Ultrasound to Predict a Pediatric Difficult Airway and Obstructive Sleep Apnea Syndrome in Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to perform the ultrasound.
Sponsor: Vidya Raman (Other)
Responsible Party: Sponsor-Investigator, Vidya Raman, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB14-00572
Record Dates: First submitted 2014-08-26; First posted 2014-08-27 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Difficult Airway; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Difficult Airway (Other): Children with a history of difficult airway intubation.
  Interventions: Procedure: Ultrasound
- Obstructive Sleep Apnea (Other): Children with a history of obstructive sleep apnea.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound to measure hyo-mental distance, tonsil size and width of the tongue.

SUMMARY:
This is a prospective study to see whether ultrasonography can predict difficult airway and/or predict obstructive sleep apnea syndrome (OSAS) in children.

ELIGIBILITY:
Inclusion Criteria:

* Children with known or suspected difficult direct laryngoscopy identified by either ENT or anesthesiologist.
* Children with difficult tracheal intubation aged 1 month - 18 years old
* Children with obstructive sleep apnea aged 1 year - 8 years old

Exclusion Criteria:

* Parent/ patient refusal to participate in study

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hyo-mental distance | intraoperative
  The distance from the hyoid bone to the mentum to predict difficult airway.

SECONDARY OUTCOMES:
Tongue width | intraoperative
  Width of the tongue between the lingual arteries.
Tonsil Size | intraoperative
  Size of tonsil (bilateral)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States